CLINICAL TRIAL: NCT01915316
Title: Measurements Of Zinc Concentration On Specimens Taken During Trans-Perineal Prostate Biopsy
Status: Completed | Type: Observational
Sponsor: ProSight (Industry)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TP001
Record Dates: First submitted 2013-07-30; First posted 2013-08-02 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prostate cancer: Men. Subjects have undergone primary and at least one secondary prostate biopsy with negative diagnostics. Elevated PSA (Prostate Specific Antigen), typically above 10 ng/mL.
  Interventions: Other: prostate biopsy

INTERVENTIONS:
Other: prostate biopsy — Measurements of Zinc concentration along fresh Specimens taken during Trans-Perineal saturated repeat Prostate Biopsy before Specimens are sent to Pathology.

SUMMARY:
The purposes of this study are to: i) confirm and improve the accuracy of the correlation between levels of Zinc in prostate tissue and the grade of prostate cancer in that tissue as determined through pathology; and ii) determine the levels of zinc in prostate tissue declared as non-cancerous by pathology and located in the vicinity of tissue declared as cancerous by pathology, and verify that the Zinc levels for the declared non-cancerous tissue are lower (statistically significantly) than the levels for benign tissue not in the vicinity of cancerous tissue.

ELIGIBILITY:
Inclusion Criteria:

* Elevated PSA, >10ng/mL
* Subject underwent primary and at least one secondary (repeat) prostate biopsy with negative diagnosis
* Subject directed at saturated trans-perineal biopsy

Exclusion Criteria:

* Subject was under Zn supplement nutrition treatment

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men. Primary biopsy and at least one secondary (repeat) biopsy diagnosed negative. Elevated PSA, >10ng/mL. Subject directed at saturated trans-perineal biopsy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Verify the existence of correlation between low levels of Zinc concentration in a biopsy specimen and the prostate cancer grade for that specimen determined by pathology. | Zinc measurements on biopsy specimens are performed during the biopsy session; pathology classification is typically performed within 2-4 weeks.

SECONDARY OUTCOMES:
Verify that the levels of zinc in non-cancerous specimens located in the vicinity of a specimen declared as cancerous by pathology are lower (statistically significantly) than the levels for benign specimens not in the vicinity of the cancerous specimen. | Time frame for pathology: within 2-4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Haim Matzkin, Prof., Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel